CLINICAL TRIAL: NCT00297401
Title: The Effect of Protein Kinase C Inhibition on Renal and Peripheral Hemodynamic Function in Patients With Type 1 Diabetes Mellitus
Brief Title: Renal and Peripheral Hemodynamic Function in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chromaderm, Inc. (Industry)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8023; B7A-CA-S003
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — ruboxistaurin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ruboxistaurin
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ruboxistaurin — 32 mg, QD, PO, up to 8 weeks
  Other Names: Arxxant; LY333531
  Arms: 1
Drug: placebo — QD, PO, up to 8 weeks
  Arms: 2

SUMMARY:
Protein kinase C (PKC), an enzyme in the body, has been implicated in the process of diabetic microvascular complications. The purpose of this study will be to evaluate the renal hemodynamic and peripheral vascular effects of PKC inhibition with ruboxistaurin mesylate (an inhibitor of PKC) in patients with Type 1 diabetes mellitus and evidence of early nephropathy. In this pilot study, 21 patients with type 1 diabetes were planned to be randomized to LY333531 or placebo in a 2:1 fashion, after an initial period of testing. After 8 weeks of study drug, patients were retested.

DETAILED DESCRIPTION:
This is a pilot study with 3 parts. Twenty-one patients with type 1 diabetes will be randomized to LY333531 or placebo in a 2:1 fashion. Each patient will be studied on four occasions, while euglycemic and while hyperglycemic without PKC inhibition and while euglycemic and hyperglycemic after an eight-week period of PKC inhibition.

Study Part 1: The impact of PKC inhibition on the renal and peripheral hemodynamic response to hyperglycemia On the evening prior to the first study day, the study participants will be admitted to an in-patient research facility with overnight plasma glucose levels maintained at 4-6 mmol/L using a modified glucose clamp technique. The next day, baseline measures of endothelial function and vascular compliance, mean arterial pressure (MAP), and renal function, including glomerular filtration rate (GFR), effective renal plasma flow (ERPF), renal blood flow (RBF), filtration fraction (FF) and renal vascular resistance (RVR) will be obtained using inulin and para-aminohippurate. In all diabetic subjects, euglycemia or hyperglycemia will be maintained by modified overnight glucose clamping techniques. During the second day of the study, capillary blood glucose will be maintained at 9-11 mmol/l overnight, and the renal and peripheral vascular hemodynamic measurements will be repeated the following day. The subjects will then be given the PKC-inhibitor LY333531 (or placebo) for 6 weeks, after which the study will be repeated. The first dose of LY333531 will be taken at 0800 hrs the day after the completion of Study 1 The dose will consist of 32 mg PO OD. Study participants will monitor their capillary blood glucose levels on a four times daily schedule.

Study Part 2: The impact of PKC inhibition on the response to Ang II On the evening prior to the first study day, the study participants will be admitted to an in-patient research facility with overnight plasma glucose levels maintained at 4-6 mmol/L using a modified glucose clamp technique. The next day, baseline measures of renal function, including GFR, ERPF, RBF, FF and RVR will be obtained. Graded Ang II infusion will be administered, and the response of MAP, GFR, RPF, RBF, FF and RVR will be measured. The subjects will then be given the PKC-inhibitor LY333531 (or placebo) for 8 weeks, as previously described, after which the study will be repeated.

Study Part 3: The impact of PKC inhibition on proteinuria . Subjects will collect a 24 hour urine sample for protein / albumin excretion. They will subsequently be randomized to receive either the PKC inhibitor LY333531 or placebo, using a table of random numbers. After 8 weeks treatment, the 24 hour urine sample will again be collected.

ELIGIBILITY:
Inclusion Criteria:

* have type 1 diabetes mellitus
* hemoglobin A1C between 6 and 10%
* have evidence of early diabetic renal disease as determined by creatinine clearance more than 80 ml/minute, urine albumin to creatinine ratio of more than 3.0 and urinary albumin levels consistent with the diagnosis of diabetic nephropathy (more than 20 mg/mmol for men and more than 28 mg/mmol for women)
* are without language barrier, cooperative, expected to return for all follow-up visits, and who give informed consent before entering the study's randomization phase and after being informed of the study medications and procedures.

Exclusion Criteria:

* Have poorly controlled diabetes, chronic liver disease, clinical jaundice, and/or elevation of liver-related laboratory results, have chronic renal failure on dialysis, have received a kidney transplant or have a moderate to severe kidney disease, have previous history of myocardial infarction, stroke, claudication or amputation, have cancer and are currently receiving chemotherapy or plan to receive chemotherapy in the next 6 months and woman of childbearing potential despite actively practicing birth control by using a medically accepted device or therapy.
* are being treated or intending to start treatment during the trial with excluded drugs: topical or oral carbonic anhydrase inhibitors and require more than 2 weeks of treatment with drugs known to strongly inhibit cytochrome P450 3A4 (CYP3A4), including but not limited to, delavirdine, fluconazole, itraconazole, indinavir, ketoconazole mibefradil, nelfinavir, ritonavir, and saquinavir.
* consume alcohol, tobacco and nicotine products within 48 hours before the study and have any condition that, in the investigator's opinion, would preclude meaningful participation in the study, including, but not limited to, abnormal laboratory values the investigator considers clinically significant, patients who are poor medical or psychiatric risks for treatment with an investigational drug, patients who are unlikely to complete the study.
* suspected or proven to have a kidney disease other than diabetic related albuminuria and/or renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary outcomes will be the change in proteinuria, pre- and post-treatment with ruboxistaurin. | Baseline and 8 weeks
Change in the renal and peripheral pressor response to hyperglycemia pre and post treatment with ruboxistaurin | Baseline and 8 weeks
Change in the renal and peripheral pressor response to Angiotensin II pre and post-treatment with ruboxistaurin. | Baseline and 8 weeks

SECONDARY OUTCOMES:
Secondary analyses will consist of the change in endothelial function and vascular compliance pre- and post-treatment with ruboxistaurin. | Baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karl Beutner, Study Director — Chromaderm, Inc.
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physcian., Toronto, Ontario, Canada

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com